CLINICAL TRIAL: NCT02920229
Title: 68Ga-PSMA, N,N'-Bis(2-hydroxybenzyl)Ethylenediamine-N,N'-Diacetic Acid (HBED)-PET/CT in the Evaluation of the Biochemical Relapse in Patients With a History of Prostate Cancer Radically Treated
Brief Title: 68Ga-PSMA HBED-PET/CT in the Evaluation of the Biochemical Relapse in Patients With a History of Prostate Cancer Radically Treated
Acronym: GaPSMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRST185.02; 2015-003397-33 (EudraCT Number)
Record Dates: First submitted 2016-04-11; First posted 2016-09-30 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: 68Ga-PSMA HBED-PET/CT; Prostate Cancer
Keywords: 68Ga-PSMA; HBED-PET/CT; biochemical relapse; prostate cancer; radically treated
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga- PSMA PET/CT (Experimental): 100-200 MBq of 68Ga-PSMA will be injected intravenously prior to perform the PET/CT
  Interventions: Drug: 68Ga- PSMA

INTERVENTIONS:
Drug: 68Ga- PSMA — 100-200 MBq of 68Ga-PSMA will be injected intravenously prior to perform the PET/CT

SUMMARY:
Single-center, prospective, diagnostic trial in radically treated patients with biochemical recurrence of prostate cancer. Patients with radically treated prostate cancer with biochemical relapse and negativity of all traditional morphological and functional imaging (transrectal ultrasound, bone scan, 18F-FMC PET/CT, CT/MRI) or doubtful imaging of 2-deoxy-2-[fluorine-18] (18F)-fluoromethylcholine (FMC) PET/CT will receive a Gallio-68 (68Ga)- Prostate Specific Membrane Antigen (PSMA) Positron Emission Tomography (PET)/Computed Tomography (CT) scan.

DETAILED DESCRIPTION:
Single-center, prospective, diagnostic trial. The primary objective of this study is to evaluate the sensitivity of 68Ga-PSMA PET /CT defined as the ratio between the number of 68Ga-PSMA PET /CT positive patients and the number of prostate cancer patients with biochemical relapse and negative standard imaging.

The secondary objectives are:

* Sensitivity for different Prostatic Specific Antigen (PSA) values (ranges)
* Sensitivity for different lesion sites
* Treatment response assessment with a second PET
* False positives detection during Follow Up (FUP) (with other standard methods and eventually optional biopsy) for patient without any treatment
* safety 67 evaluable patients will be injected with 100-200 megabecquerel (MBq) 68Ga-PSMA intravenously

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed prostate cancer
2. Male, aged >18 years.
3. Radical treatment for prostate cancer (radiotherapy or surgery)
4. 18F-FMC PET/CT negative or doubtful
5. Negativity of all the other traditional morphological and functional imaging (transrectal ultrasound, bone scan, CT/MRI)
6. Patients with PSA progression defined as PSA ≥ 1,0 ng/mL and/or PSA rising defined as 2 subsequent values showing PSA increase at least 1 week apart.
7. Male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
8. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. No hormonotherapy in the last 6 months
2. No radiotherapy in the last 6 months.
3. Patients with PSA < 1.0 ng/ml
4. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Study Agent.
6. Medical or psychological conditions that would not permit the subject to complete to sign informed consent

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1230 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
the ratio between the number of 68Ga-PSMA PET/CT positive patients and the number of prostate cancer patients with biochemical relapse and negative standard imaging | up to 24 months
  the ratio between the number of 68Ga-PSMA PET/CT positive patients and the number of prostate cancer patients with biochemical relapse and negative standard imaging

SECONDARY OUTCOMES:
Sensitivity for different PSA values (ranges) | up to 24 months
  Sensitivity of 68Ga- PSMA PET/CT for different PSA values (ranges)
Sensitivity for different lesion sites | up to 24 months
  Sensitivity of 68Ga- PSMA PET/CT for different lesion sites
PSA decrease: the receiver operating characteristic (ROC) curves generated by plotting sensitivity versus 1-specificity. Youden's index will be used for determining cut-off value between pos and neg 68Ga-PSMA PET/CT findings | up to 24 months
  for patients that will start an anticancer treatment: evaluate the predictive role of 68Ga- PSMA PET/CT on early response to therapy (hormonotherapy, abiraterone, enzalutamide) taking PSA decrease as a reference.
Evaluation of the concordance between 68Ga- PSMA PET/CT and PET/CT or the others standard methods, performed by the Cohen's kappa coefficient. | up to 24 months
  for patient without any treatment: evaluate the concordance between 68Ga- PSMA PET/CT and other standard methods and eventually optional biopsy
number of treated patients experiencing grade 1 to 4 adverse events | up to 24 months
  number of treated patients undergoing grade 1 to 4 adverse events evaluated according to CTCAE v.4.0
percentage of treated patients experiencing grade 1 to 4 adverse events | up to 24 months
  percentage of treated patients experiencing grade 1 to 4 adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Federica Matteucci, MD, Principal Investigator — IRST IRCCS, Meldola (FC)
Locations (1):
- Irst Irccs, Meldola, FC, Italy

IPD SHARING:
Plan to Share IPD: Undecided
undecided